CLINICAL TRIAL: NCT01619514
Title: Uncovering Potential Breast Cancer Biomarkers Amp; Possible Drug Targets Using Advanced Quantitative Mass Spectrometry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/00106
Record Dates: First submitted 2012-04-02; First posted 2012-06-14 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the use of advanced quantitative mass spectometry (Super SILAC) as a discovery platform to uncover novel protein biomarkers in tumor and to compare the protein profile between different subtypes of breast cancer (ER positive, HER2 positive, triple negative). A maximum of 100 breast tumor specimens will be obtained from the NUHS Tissue repository, comprising approximately equal proportion of ER positive, HER2 positive, and triple negative tumors. Samples will be analyzed using advanced Mass Spectrometry (Super SILAC) as a discovery platform to identify novel protein biomarkers that may be important in cancer. DNA and RNA will also be extracted from tumor samples for correlative analysis with the proteomics data. Genomics and proteomics data will be correlated with clinical data including treatment response and survival data. Importance of proposed research to science or medicine:Identification of tumor biomarkers may allow better prognostication, follow-up, and selection of treatment for cancer patients in the future. Potential benefits and risks: No direct benefit to the patient. Risk to the subjects is minimal as there is no direct patient contact, and analysis is done on previously donated tumor samples. Patients have previously provided consent to donate their samples for research into the NUHS Tissue Repository.

Novel tumor biomarkers that determine tumor biology, including prognosis and treatment sensitivity, may be detectable using the novel advanced quantitative mass spectromy method (Super SILAC). Different subtypes of breast cancers will have different proteomic profiles analyzed using super SILAC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tumor specimens that have been stored in the NUHS tissue repository will be retrieved
Sampling Method: Probability Sample
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the use of advanced quantitative mass spectometry (Super SILAC) as a discovery platform to uncover novel protein biomarkers in tumor
  SILAC is a method of advanced quantitative mass spectometry that allows whole proteome analysis as comprehensively as transcriptome analysis. It allows quantification of whole-proteome, measure post-translational modifications and map complete interactome of a protein. Super-SILAC, an improvement of the SILAC method, enables the comparison of the amounts of hundreds or thousands of proteins from a particular tissue between different patients. This technology may enable the discovery of novel tumor protein markers that may be important in tumor progression and treatment response.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationa University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Geiger T, Cox J, Ostasiewicz P, Wisniewski JR, Mann M. Super-SILAC mix for quantitative proteomics of human tumor tissue. Nat Methods. 2010 May;7(5):383-5. doi: 10.1038/nmeth.1446. Epub 2010 Apr 4. PMID 20364148
- [Background] Neubert TA, Tempst P. Super-SILAC for tumors and tissues. Nat Methods. 2010 May;7(5):361-2. doi: 10.1038/nmeth0510-361. No abstract available. PMID 20431548